CLINICAL TRIAL: NCT05467709
Title: A Phase 1, Open-Label, Fixed-Sequence, Drug-Drug Interaction Study To Evaluate The Effect Of Multiple Doses of CTP-543 On The Pharmacokinetics Of Single Doses of Midazolam In Healthy Subjects
Brief Title: Study To Evaluate The Effect Of Multiple Doses of CTP-543 On The Pharmacokinetics Of Single Doses of Midazolam In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP543.1012
Record Dates: First submitted 2022-06-30; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Health Volunteers
Keywords: CTP-543
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTP-543 (Experimental): Subjects will receive a single 2 mg dose of midazolam on Day 1. Starting on Day 3, 12 mg dose of CTP-543 will be administered (q12 hrs) for 14 consecutive days (up to Day 16). On Day 16, subjects will be co-administered a single 2 mg midazolam dose along with the morning dose of CTP-543. The second dose of CTP-543 will be administered as scheduled on Day 16.
  Interventions: Drug: Midazolam; Drug: CTP-543

INTERVENTIONS:
Drug: Midazolam — 2 mg Day 1 and Day 16
Drug: CTP-543 — 12 mg q12 hour for 14 consecutive days starting on Day 3

SUMMARY:
This is a single center, Phase 1, open-label, fixed-sequence, drug-drug interaction study to determine the effect of CTP-543 on the pharmacokinetics (PK) of midazolam in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, aged 18-60
* Non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at screening
* If of reproductive age, willing and able to use a medically highly effective form of birth control 4 weeks prior to first dose, during the study and for 30 days following last dose of study medication
* Capable of giving informed consent and complying with study procedures

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease
* History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing
* Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
* History of prolonged QT syndrome or a QTc interval with Fridericia's correction (QTcF) > 450 msec for males or QTcF > 470 msec for females at screening visit or prior to the first dosing
* Abnormal liver function at screening
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study drug
* Positive results for coronavirus infection (COVID-19) at screening or check-in
* Positive drug or alcohol results at screening or check-in
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* Participation in another clinical study within 30 days prior to, and 30 days after the first dosing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 14, 15, 16, Discharge (Day 17)
  Maximum observed concentration
Tmax | Day 14, 15, 16, Discharge (Day 17)
  Time to reach maximum observed concentration
AUC0-inf | Day 14, 15, 16, Discharge (Day 17)
  Area under the concentration-time curve from time 0 extrapolated to infinity
AUC0-t | Day 14, 15, 16, Discharge (Day 17)
  Area under the concentration-time curve from time 0 to the time of the last observed/measured non-zero concentration
λz | Day 14, 15, 16, Discharge (Day 17)
  Terminal elimination rate constant
t1/2 | Day 14, 15, 16, Discharge (Day 17)
  Apparent terminal half-life
CL/F | Day 1, 2, 16, Discharge (Day 17)
  Apparent total plasma clearance (Midazolam only)
Vz/F | Day 1, 2, 16, Discharge (Day 17)
  Apparent volume of distribution (Midazolam only)

SECONDARY OUTCOMES:
Assessment of Safety and Tolerability following administration of CTP-543 | Screening (within 21 days prior to Day 1) through follow-up (approximately 7 days after last study drug administration)
  Number of adverse events, including abnormal clinical laboratory findings, abnormal physical examinations, abnormal ECGs and abnormal vital signs tabulated for each subject

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, LLC, Miami, Florida, United States